CLINICAL TRIAL: NCT07157995
Title: Building Active Living and Addressing Needs for Caregiver Empowerment (BALANCE) Study - Phase 4 of Designed With You
Brief Title: Phase 4 of Designed With You
Acronym: BALANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00388844
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Disability Physical
Keywords: Caregivers; Disability; Sensory Disability; Mobility Disability

STUDY DESIGN:
Intervention Model Description: feasibility study of the BALANCE intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance Intervention (Other): Participants will receive the intervention. BALANCE is a feasibility study of the BALANCE intervention that is testing feasibility and acceptability of a intervention that includes individual and group sessions with a caregiver navigator. The focus of the intervention is the unmet needs of caregivers with disabilities.
  Interventions: Behavioral: BALANCE Building Active LIving and Addressing Needs for Caregiver Empowerment

INTERVENTIONS:
Behavioral: BALANCE Building Active LIving and Addressing Needs for Caregiver Empowerment — The Balance intervention will include individual visits by a Caregiver Navigator and group sessions with other participants, led by the caregiver navigator. The focus will be on future planning, resources for unmet needs and support and socialization.

SUMMARY:
The purpose of this study is to provide evaluate the feasibility of a structured 8-10-week, multi-component intervention that integrates individualized resource navigation, personalized self-care planning, emergency and end of life (EOL) preparedness, and peer support to improve the well-being, resource access and social connectedness of caregivers with disabilities. For this study we are interested in caregivers over the age of 18 who have some form (e.g. mobility or sensory) disability and are caring for a person with a disability and/or a chronic illness.

DETAILED DESCRIPTION:
The BALANCE is a feasibility study of the BALANCE intervention and will be delivered over 8-10 weeks. The proposed study is a Phase 1 feasibility trial designed to assess the feasibility and acceptability of a novel intervention aimed at [briefly describe intervention]. The primary objectives are to evaluate the practicality of implementing the intervention, participant engagement, and the appropriateness of study procedures.

Given the early-stage nature of this research, a control group is not required. Phase 1 feasibility studies are not intended to assess efficacy or comparative outcomes, but rather to refine the intervention and study logistics. According to guidance from the Office of Research Integrity (ORI), "Phase I trials are feasibility trials focused on developing and pretesting the acceptability, feasibility, and safety of the intervention components of Balance. "No control condition is needed."14 This approach aligns with best practices in early intervention development and allows for iterative refinement before proceeding to more rigorous testing in later phases (e.g., randomized controlled trials).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older,
* Community dwelling in the state of Maryland,
* Self report of physical or sensory disability and
* self-report of serving as a family caregiver for a person for at least 10 hours/week.

Exclusion Criteria:

* have a terminal diagnosis (<1 year expected survival), and
* > severe cognitive impairment (5-7 errors) based on the Short Portable Mental Status Questionnaire (SPMQ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Baseline and post intervention at approximately 10 weeks
  Measurement of perceived stress. Scores can range from 0 to 40, with higher scores indicating worse levels of perceived stress.
Caregiver Burden Short Form | Baseline and post intervention at approximately 10 weeks
  Measure to address burdensome activities related to care giving experiences. Total score ranges from 0-48 wit higher scores indicating greater caregiver burden.
Depressive Symptoms (PHQ-9) | Baseline and post intervention at approximately 10 weeks
  Measure of depressive symptoms. Score range 0-27, higher values represent more depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Janiece Taylor, PhD, RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No